CLINICAL TRIAL: NCT02367976
Title: A Phase III Study to Research the Efficacy and Safety on Prouk for ST Elevated Mycadial Infarction Patients in China
Brief Title: Efficacy and Safety on Prouk for STEMI Patients in China
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suzhou RxD Biopharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012L01494
Record Dates: First submitted 2015-01-15; First posted 2015-02-20 (Estimated); Last update posted 2015-02-25 (Estimated); Status verified 2015-02

CONDITIONS: STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- rhprouk (Experimental): rhprouk to be administrated in 60 minutes.
  Interventions: Drug: rhprouk
- controlled (No Intervention): The controlled arm patients will be administrated in 90 minutes after randomized.

INTERVENTIONS:
Drug: rhprouk — rh-prouk will be administrated within 60 minutes after the patients eligibility confirmed
  Other Names: Controlled
  Arms: rhprouk

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of rh-prouk as pharmacoinvasive therapy on those ST Elevated Myocardial Infarctions patients, it is designed as a multicenter, active controlled, single blinded study. The primary endpoint is to assess the coronary recanalization 90 minutes after thrombolysis. The secondary endpoint is to evaluate the mortality rate at day 30.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the efficacy and safety of rh-prouk as pharmacoinvasive therapy on those ST Elevated Myocardial Infarctions patients, it is designed as a multicenter, active controlled, single blinded study. The primary endpoint is to assess percentage of patients achieve the coronary recanalization 90 minutes after thrombolysis. The secondary endpoint is to evaluate the mortality rate at day 30.

ELIGIBILITY:
Inclusion Criteria:

* Chest pain > 30 minutes, while <12 hours
* Expected PCI related delayed time > 60 minutes, OR Door To Balloon time >90 minutes
* ECG confirmed STEMI.
* Age: 18--75 years old
* Weight <=85Kg
* Consent to participate in this study

Exclusion Criteria

* Evidence of cardiac rupture;
* ECG: new left bundle branch block;
* Thrombolysis contradictions
* Any history of central nervous system damage (i.e. neoplasm, aneurysm, intracranial or spinal surgery) or recent trauma to the head or cranium (i.e. < 3 months);
* Active bleeding or known bleeding disorder.
* Recent administration of any i.v. or s.c. anticoagulation within 12 hours includingunfractionated heparin, enoxaparin and/or bivalirudin or current use of oral anticoagulation(warfarin or coumadin);
* Uncontrolled hypertension, defined as a single blood pressure measurement ≥ 180/110 mm Hg (systolic BP ≥ 180 mm Hg and/or diastolic BP ≥ 110 mm Hg) prior to randomisation;
* Major surgery, biopsy of a parenchymal organ, or significant trauma within the past 2 months (this includes any trauma associated with the current myocardial infarction); Prolonged or traumatic cardiopulmonary resuscitation (> 10 minutes) within the past 2 Weeks Major surgery pending in the following 30 days;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
To compare the percentage of STEMI patients achieving the recanalization of Coronary between the two arms | 90 minutes after administrative of active/comparator

CONTACTS AND LOCATIONS:
Overall Officials: Weiqun Shen, MD/PhD, Study Director — Suzhou RxD Biopharma
Locations (1):
- Shenyang Northern Hospital, Shenyang, Liaoning, China